CLINICAL TRIAL: NCT00300118
Title: Double-blind, Double-dummy, Randomized, Multicentre Study to Compare the Efficacy and Safety of Oral Budesonide (9 mg) and Oral Mesalazine (4.5 g) in Moderately Active Crohn's Disease Patients
Brief Title: Oral Budesonide vs. Oral Mesalazine in Active Crohn's Disease (CD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUC-52/CDA; 2004-001213-34
Record Dates: First submitted 2006-03-07; First posted 2006-03-08 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Budesonide; Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: budesonide
- B (Active Comparator)
  Interventions: Drug: mesalazine

INTERVENTIONS:
Drug: budesonide — 9 mg
  Arms: A
Drug: mesalazine — 4.5 g
  Arms: B

SUMMARY:
The purpose of this study is to determine whether mesalazine or budesonide is more active in the treatment of active Crohn's disease.

DETAILED DESCRIPTION:
Crohn's disease is often treated with glucocorticoids or mesalazine. Both drugs are indicated for active Crohn's disease. Treatment with mesalazine is indicated for the treatment of mildly to moderately active Crohn's disease. Budesonide 9 mg/day or mesalazine 4.5 g/day are better than lower doses.

So far only one trial compares the efficacy and safety of budesonide and 5-ASA. The result of this trial is that budesonide is more effective in inducing remission than mesalazine. The primary objective of this trial is to confirm this result for other presentations of budesonide and mesalazine; i.e. Budenofalk® capsules (9 mg/day) and Salofalk® tablets (Eudragit-L-coated oral mesalazine; 4.5 g/day) in moderately active Crohn's disease. Mesalazine is used in this trial as a comparator.

ELIGIBILITY:
Inclusion Criteria (main):

* Symptoms of Crohn's disease since at least 3 months; diagnosis confirmed by endoscopic and histological, or endoscopic and radiological criteria [endoscopy not older than 12 months or if older, then clinical signs (e.g. pain localization, pain intensity, blood in stool) and behaviour (according to Vienna classification) should be unchanged compared to former episodes]
* Localisation of CD either in terminal ileum, ascending colon or ileocolitis
* Active phase of disease (200 < CDAI < 400)

Exclusion Criteria (main):

* Known Crohn's lesion in the upper GI-tract (up to and including the jejunum) with present symptoms
* CD in the rectum currently present
* Short bowel syndrome
* Septic complications
* Baseline stool positive for germs causing bowel disease
* Abscess, perforation or active fistulas
* Ileostomy or colostomy
* Resection of more than 50 cm of the ileum
* Bowel surgery within the last 3 months
* Immediate surgery required
* Clinical signs of stricturing disease
* Subileus within the last 6 months
* Suspicion of ileus, subileus or corresponding symptomatology
* Contra-indications, special warnings and precautions mentioned in SmPC
* Treatment with immunosuppressants, cytostatics, 6-TG, methotrexate, or cyclosporine within the last 3 months; in case of treatment with azathioprine or 6-MP the drugs have to be used for maintenance of remission only and dosage has to be unchanged within the last 3 months before baseline visit and during the study
* Treatment with ketoconazole, ciprofloxacin or other CYP3A inhibitors within the last month before baseline visit
* Treatment with anti-TNF-a therapy within 6 months before baseline visit
* Conventional steroids (iv, po, rectal) within 2 weeks before the study
* > 6 mg/d budesonide po or > 3 g/d mesalazine po within 2 weeks before the study
* Patients known to be steroid-refractory or steroid-dependent from former CD episodes
* Treatment of study disease with oral antibiotics (e.g., metronidazole) within the last 2 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2004-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Rate of remission

SECONDARY OUTCOMES:
Response to treatment
Time to response
Time to remission
PGA
QoL

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Tromm, Professor, Principal Investigator — Ev. Krankenhaus Hattingen GmbH
Locations (1):
- Ev. Krankenhaus Hattingen GmbH, Hattingen, Germany

REFERENCES:
- [Result] Tromm A, Bunganic I, Tomsova E, Tulassay Z, Lukas M, Kykal J, Batovsky M, Fixa B, Gabalec L, Safadi R, Kramm HJ, Altorjay I, Lohr H, Koutroubakis I, Bar-Meir S, Stimac D, Schaffeler E, Glasmacher C, Dilger K, Mohrbacher R, Greinwald R; International Budenofalk Study Group. Budesonide 9 mg is at least as effective as mesalamine 4.5 g in patients with mildly to moderately active Crohn's disease. Gastroenterology. 2011 Feb;140(2):425-434.e1; quiz e13-4. doi: 10.1053/j.gastro.2010.11.004. Epub 2010 Nov 9. PMID 21070781